CLINICAL TRIAL: NCT03755479
Title: Evaluation of Minimed 670G Hybrid Closed Loop System On-Boarding Protocol, for Patients With Type 1 Diabetes on Multiple Daily Insulin Injection Therapy
Brief Title: Evaluation of Minimed 670G in T1D Patients on Multiple Daily Injection
Status: Completed | Type: Observational
Sponsor: Sidra Medicine (Other)
Responsible Party: Principal Investigator, Goran Petrovski, Goran Petrovski, MD PhD, Sidra Medicine
Other Study IDs: 1810033883
Record Dates: First submitted 2018-11-25; First posted 2018-11-28 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus Type 1; Insulin Pump; Hybrid closed Loop System; Minimed 670G
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Single Arm Group: Patient on multiple daily injections will start Hybrid Closed Loop System Insulin Pump Minimed 670G
  Interventions: Device: Hybrid Closed Loop Insulin Pump Minimed 670G

INTERVENTIONS:
Device: Hybrid Closed Loop Insulin Pump Minimed 670G — Five Day Group Education on Minimed 670G

SUMMARY:
Introduction. Sensor Augmented Pump has demonstrated superiority over insulin pump and Multiple Daily Injection (MDI) in achieving optimal glucose control and can improve quality of life in Type 1 Diabetes (T1D) patients. Hybrid closed loop (HCL) insulin pump Minimed 670G is a FDA approved device and European Conformity (CE) mark with SmartGuard technology and closed loop algorithm, which will allow the patients to improve their diabetes management. Hybrid closed loop insulin pump Minimed 670G monitors glucose in the subcutaneous tissues and automatically adjusts the delivery of rapid acting insulin as basal rate based on the user's glucose reading. SmartGuard technology in insulin pump, based on user's sensor glucose values can predict when glucose is approaching low levels, 30 minutes in advance and automatically stop insulin delivery. When user's glucose levels recover, SmartGuard will automatically resume insulin delivery. CareLink is personal software, which downloads the data from insulin pump, glucose sensor and glucometer to visualize diabetes information with charts, statistics and events that help patient and health provider to identify and understand patterns and trends The objective of this study is to assess structured group education on boarding protocol of the HCL Minimed 670 G in achieving glucose control of patients on MDI.

Methods. This study is a single-arm, single-center, clinical investigation in subjects with type 1 diabetes on HCL insulin pump (Minimed 670G) in a period of 3 months. A total of 30 subjects (age 6 - 17) will be enrolled in order to reach 26 subjects who will complete the HCL study. The investigators will start the clinical process for initiating an insulin pump, which is typically done with pre-pump classes. HbA1c, derived from CGM will be performed at baseline and 3 months during the study. The following parameters will be analyzed: % patients achieving Time in Range (TIR) > 67% from 70 mg/dl to 180 mg/dl; % patients achieving TIR <3%, below time in range (<70 mg/dl) and % patients achieving both TIR > 67% and <3% time below Range. Collection of demographics and medical history, data for diabetes devices (eg meters, sensors, pumps) and brief clinical physical exam including vital signs and skin assessment will be obtained via Hospital Electronic Medical File (Cerner Millennium, North Kansas City, US) and will be kept as electronic data on a separate research server.

DETAILED DESCRIPTION:
This study is a single-arm, single-center, clinical investigation in subjects with Type 1 Diabetes (T1D) on Hybrid Closed Loop (HCL) insulin pump Minimed 670G in a period of 3 months. A total of 30 subjects (age 6 - 17) will be enrolled in order to reach 26 subjects who will complete the HCL study.

After reviewing the patient's eligibility and interest, the investigators will obtain informed consent and assent as appropriate. The investigators will start the clinical process for initiating an insulin pump, which is typically done with pre-pump classes. HbA1c, derived from Continuous Glucose Monitoring (CGM) device will be analyzed at baseline and 3 months during the study.

Collection of demographics and medical history, data for diabetes devices (eg meters, sensors, pumps) and brief clinical physical exam including vital signs and skin assessment will be obtained via Hospital Electronic Medical File (Cerner Millennium, North Kansas City) and will be kept as electronic data on a separate research server.

Base line assessment

The main variables checked at baseline:

* Age
* Duration of diabetes
* Total daily insulin (TDI) dose
* HbA1c, derived from CGM device

Recruitment process All patients will be recruited during the regular clinic visits at Diabetes Clinics at Sidra Medicine in Doha. The Principal investigator will evaluate the patient if meets the inclusion criteria during the regular clinic visits. A research assistant will take patient and family in other room to explain the study protocol and give patient information. Parents and patients can ask questions about the study. After the explanation of the study protocol, if parents and child agree to participate, they can sign the documents for including in the study. Parents can also take the documents home to consider the possible inclusion in the study. They can also talk to principal investigator before including the child in the study. If parents agree to be a part of the study, they can call research assistant to include the child in the study. The research assistant will arrange a separate meeting to start the process.

Run in period The 2-week run-in period will be used for education and training for the new devices.

Week 1: Pump school (Sunday to Thursday) A group session of 2-3 patients/families will be performed to allow subject to become familiar with new insulin pump. Five sessions in a row (each two hours) will be performed during a week.

Glucose sensor (Suspend before low and suspend on low will be off) will be started on the first day (Same protocol which is currently used in Sidra Medicine).

Topics and education Sunday: Basal Bolus Concept; Operational modes of the pump; Understanding the pump; Pump buttons; Glucose readings; Reading the display; Sensor alerts and alarms; How to insert a sensor; Pump menus Monday: Carelink personal; Battery change; Setting date and time; Basal rates; Pump suspend; Bolus wizard, Bayer Contour Next Link 2.4 Tuesday: Infusion set change; Alarms and alerts; Suspend before low and Suspend of low; Advanced carbs counting Wednesday: Temporary basal; Emergency kit; Low blood sugar; High Blood Sugar; Sick day's management for pump; Diabetic Ketoacidosis (DKA)' Blood glucose Blood ketones; Exercise; Travel Thursday: Auto Mode; Using Auto Mode for the first time Checking Auto Mode Readiness; sensor graph in Auto Mode' Using pump in Auto Mode; Entering a Blood Glucose value in Auto Mode; Suspending and Resuming Delivery in Auto Mode Evaluation Check List; Pump Care; Setting the pump; Sensor start by patient The sensor will be started the first day for teaching and observational purposes only. CareLink account creation and sharing of access is mandatory in the first week.

Week 2: Pump start (Sunday to Sunday) Sensor Augmented Pump will be initiated with both Smart Guard and HCL turned off, to allow the investigators, subjects and device to get more information before starting the HCL. This week will be used as a warm up period for Auto Mode.

Study Period 3 Months Following the two week run-in period using the Minimed 670G, Auto Mode will be activated and all subjects will participate in a 3-month study period.

The patient/family will upload data into the CareLink system and the data will be reviewed by a member of the clinical team. Adjustments to system settings will be suggested to the family as clinically appropriate.

Visit 1- Day 1 In-Clinic visit. Insulin pump will be started in Auto mode. Carelink download for initial pump settings. HbA1c will be obtained.

Visit 2- Day 3 Remote visit. Download pump at home, phone call to patient. Check the Auto Mode, pump settings and fine tune.

Visit 3- Day 7 In-Clinic visit. Download pump. Check the Auto Mode, pump settings and fine tune. Visit 4- Day 14 Remote visit. Download pump at home, phone call the patient. Check the Auto Mode, pump settings and fine tune.

Visit 5- Day 28 In-Clinic visit. Month 1 Download pump. Check the Auto Mode, pump settings and fine tune. Visit 6- Day 42 Remote visit. Download pump at home, phone call to patient. Check the Auto Mode, pump settings and fine tune.

Visit 7- Day 84 In-Clinic visit. Month 3 Download pump. HbA1c will be obtained.

Data Analysis The analysis of the main endpoint 3 month Time in Range, post intervention will be tested by the paired student t-test or paired Wilcoxon test, in case of non-normality of the end point. Evident outliers will be excluded from the main analysis but data on the complete analysis will be provided as well.

The different continuous baseline values will be checked for normality of distribution using the mean-median comparison, skewness and kurtosis (-3 to +3), spread, Kolmogorov-Smirnow and Shapiro-Wild tests, outliers, histograms and Q-Q-plots.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Type 1 Diabetes. Diagnosis of Type 1 Diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not required.
2. HbA1c < 12.5%
3. Age 6-17 years at the initiation of the 670G system
4. Multiple Daily Injections (Basal Bolus therapy) with Total Daily Insulin use of great than 8.0 units per day over a 1 week period
5. Willing and able (access to internet from home) to download information into the Medtronic CareLink software
6. Clinically planning to and be able to start the Medtronic 670G HCL system
7. History of 3 clinic visits in the last year

Exclusion Criteria:

1. DKA in the 6 months prior to screening visit

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with Type 1 Diabetes on Multiple Daily Injections, motivated and willing to switch Hybrid Closed Loop Minimed 670G.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-11 (Actual)

PRIMARY OUTCOMES:
Achieving glucose values more than 67% in Time in Range (70-180 mg/dl) | 3 months
  Primary outcome is to achieve glucose levels more than 67% in range between 70mg and 180 mg/dl using Minimed 670G

SECONDARY OUTCOMES:
Change in HbA1c | 3 months
  Change in HbA1c levels from previous treatment (multiple daily injections) compared to Minimed 670G treatment
Glucose values above Range (>180 mg/dl) | 3 months
  Percentage of glucose values more than 180 mg/dl on Minimed 670G
Time spend in Auto Mode | 3 months
  Percentage of time in Auto Mode, where Minimed 670G automatic adjusts the basal insulin dose according glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Goran Petrovski, MD, PhD, Principal Investigator — Sidra Medicine
Locations (1):
- Sidra Medicine, Doha, Qa, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ly TT, Roy A, Grosman B, Shin J, Campbell A, Monirabbasi S, Liang B, von Eyben R, Shanmugham S, Clinton P, Buckingham BA. Day and Night Closed-Loop Control Using the Integrated Medtronic Hybrid Closed-Loop System in Type 1 Diabetes at Diabetes Camp. Diabetes Care. 2015 Jul;38(7):1205-11. doi: 10.2337/dc14-3073. Epub 2015 Jun 6. PMID 26049550
- [Background] Ly TT, Weinzimer SA, Maahs DM, Sherr JL, Roy A, Grosman B, Cantwell M, Kurtz N, Carria L, Messer L, von Eyben R, Buckingham BA. Automated hybrid closed-loop control with a proportional-integral-derivative based system in adolescents and adults with type 1 diabetes: individualizing settings for optimal performance. Pediatr Diabetes. 2017 Aug;18(5):348-355. doi: 10.1111/pedi.12399. Epub 2016 May 18. PMID 27191182
- [Background] de Bock MI, Roy A, Cooper MN, Dart JA, Berthold CL, Retterath AJ, Freeman KE, Grosman B, Kurtz N, Kaufman F, Jones TW, Davis EA. Feasibility of Outpatient 24-Hour Closed-Loop Insulin Delivery. Diabetes Care. 2015 Nov;38(11):e186-7. doi: 10.2337/dc15-1047. Epub 2015 Aug 27. No abstract available. PMID 26316630
- [Background] Bergenstal RM, Garg S, Weinzimer SA, Buckingham BA, Bode BW, Tamborlane WV, Kaufman FR. Safety of a Hybrid Closed-Loop Insulin Delivery System in Patients With Type 1 Diabetes. JAMA. 2016 Oct 4;316(13):1407-1408. doi: 10.1001/jama.2016.11708. No abstract available. PMID 27629148
- [Background] Ruiz JL, Sherr JL, Cengiz E, Carria L, Roy A, Voskanyan G, Tamborlane WV, Weinzimer SA. Effect of insulin feedback on closed-loop glucose control: a crossover study. J Diabetes Sci Technol. 2012 Sep 1;6(5):1123-30. doi: 10.1177/193229681200600517. PMID 23063039
- [Background] de Bock M, Dart J, Roy A, Davey R, Soon W, Berthold C, Retterath A, Grosman B, Kurtz N, Davis E, Jones T. Exploration of the Performance of a Hybrid Closed Loop Insulin Delivery Algorithm That Includes Insulin Delivery Limits Designed to Protect Against Hypoglycemia. J Diabetes Sci Technol. 2017 Jan;11(1):68-73. doi: 10.1177/1932296816668876. Epub 2016 Sep 25. PMID 27621143
- [Background] Bailey TS, Ahmann A, Brazg R, Christiansen M, Garg S, Watkins E, Welsh JB, Lee SW. Accuracy and acceptability of the 6-day Enlite continuous subcutaneous glucose sensor. Diabetes Technol Ther. 2014 May;16(5):277-83. doi: 10.1089/dia.2013.0222. Epub 2014 Apr 7. PMID 24758729
- [Background] Tauschmann M, Allen JM, Wilinska ME, Thabit H, Acerini CL, Dunger DB, Hovorka R. Home Use of Day-and-Night Hybrid Closed-Loop Insulin Delivery in Suboptimally Controlled Adolescents With Type 1 Diabetes: A 3-Week, Free-Living, Randomized Crossover Trial. Diabetes Care. 2016 Nov;39(11):2019-2025. doi: 10.2337/dc16-1094. Epub 2016 Sep 9. PMID 27612500